CLINICAL TRIAL: NCT05284890
Title: A Phase 1, Single-center, Open-label Study to Evaluate the Metabolism and Excretion of [14C]CC-99677 in Healthy Male Participants
Brief Title: A Study to Evaluate the Drug Levels of [14C]CC-99677 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IM046-001
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: CC-99677; Healthy Male Participants; Pharmacokinetics; Absorption; Distribution; Metabolism; Excretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-99677 (Experimental)
  Interventions: Drug: CC-99677

INTERVENTIONS:
Drug: CC-99677 — Specified dose on specified days

SUMMARY:
The purpose of the study is to characterize the absorption, distribution, metabolism and excretion (ADME) of a single oral dose of [14C] CC-99677.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants
* Body mass index of 18.0 to 33.0 kg/m^2, inclusive

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Any major surgery within 4 weeks of intervention administration
* History of any significant drug allergy

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of the drug (Cmax) for CC-99677 | Up to 15 days
Time of maximum observed plasma concentration (Tmax) for CC-99677 | Up to 15 days
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) for CC-99677 | Up to 15 days
Total radioactivity recovered in urine (UR) | Up to 15 days
Percent of total radioactivity recovered in urine (%UR) | Up to 15 days
Total radioactivity recovered in feces (FR) | Up to 15 days
Percent of total radioactivity recovered in feces (%FR) | Up to 15 days
Total radioactivity recovered in bile (BR) | Up to 15 days
Total radioactivity recovered in urine, feces, and bile combined (Rtotal) | Up to 15 days
Percent of total radioactivity recovered in all excreta (%Total) | Up to 15 days
Plasma AUC (total radioactivity (TRA))/Blood AUC (TRA) | Up to 15 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 50 days
Incidence of serious adverse events (SAEs) | Up to 50 days
Incidence of AEs leading to discontinuation | Up to 15 days
Incidence of vital sign abnormalities | Up to 15 days
Incidence of electrocardiogram (ECG) abnormalities | Up to 15 days
Incidence of physical examination abnormalities | Up to 15 days
Incidence of clinical laboratory test abnormalities | Up to 15 days
Cmax | Up to 15 days
Tmax | Up to 15 days
AUC(0-T) | Up to 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Madison, Wisconsin, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm